CLINICAL TRIAL: NCT06803602
Title: Evaluating the Efficacy of High-Intensity Focused Electromagnetic Technology in Improving the Time of Recovery of Urinary Control of Continence and Quality of Life for Post-Surgical Patients
Brief Title: HIFEM Technology for Post-Radical Prostatectomy and Post-Holmium Laser Prostate Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mitchell Humphreys, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 24-010450
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Holmium Laser Prostate Surgery; Radical Prostatectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group (Experimental): Subjects randomized to the treatment group will receive 2, 30-minute sessions, weekly for 3 weeks using the Emsella device.
  After a 1 week wash-out period, subjects still experiencing urinary leakage will have the option to continue treatment for 3 additional weeks.
  Interventions: Device: EMSELLA®
- Placebo Group (Sham Comparator): Subjects randomized to the placebo group will receive 2, 30-minute sessions, weekly for 3 weeks using a sham comparator device.
  After a 1 week wash-out period, subjects in the placebo group who are experiencing urinary leakage will be offered the opportunity to cross-over to an active treatment group for an additional 3 weeks.
  Interventions: Device: Sham Comparator Device

INTERVENTIONS:
Device: EMSELLA® — Subjects will receive 100% intensity of the EMSELLA® (BTL Industries, Marlborough, MA) High-Intensity Focused Electromagnetic (HIFEM) treatment, in a single 30-minute session, twice per week for 3 weeks.
  Arms: Treatment Group
Device: Sham Comparator Device — Subjects will be asked to sit on the EMSELLA® (BTL Industries, Marlborough, MA) treatment head which will be powered off and instead have a small remote control vibration device that will simulate active treatment, in a single 30-minute session, twice per week for 3 weeks.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of High-Intensity Focused Electromagnetic (HIFEM) technology in improving the recovery time of urinary control and quality of life for male patients after radical prostatectomy (RP) and Holmium laser prostate surgery (HoLEP).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are male
* Post-radical prostatectomy or post HoLEP
* Experiencing urinary incontinence one-month post-RP
* Have the capacity to make their own medical decisions
* Able to complete the questionnaires and visits required.

Exclusion Criteria:

* Subjects who are not male
* Not post-radical prostatectomy or post HoLEP
* Neurologic disease
* Atonic or hypofunctional bladder (bladder contractility index (BCI) < 100; BCI = pDetQmax+5Qmax)
* Status post pelvic radiation
* Past surgical history of other GU surgeries
* Gross hematuria
* Concomitant use of medications that cause muscle relaxation or inhibition
* Indwelling foley catheter at time of treatment
* Documented urine leak
* Not experiencing urinary incontinence
* Do not have the capacity to make their own medical decisions
* Unable to complete the questionnaires provided.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire Short-Form (ICIQ-SF) | Baseline, 6 weeks, 15 weeks
  The International Consultation on Incontinence Questionnaire (ICIQ-SF) is a 4-item questionnaire that assesses the frequency, amount, and impact of urinary leakage. The ICIQ-SF has a scoring range of 0-21, with higher scores indicating more severe symptoms.
Pad weight test | Baseline, 6 weeks, 15 weeks
  For the pad weight test, subjects will be provided with a small scale and asked to measure the weight of their pad before and after wearing for 24 hours.

SECONDARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Baseline, 6 weeks, 15 weeks
  The International Prostate Symptom Score (IPSS) is a 7-item questionnaire used to assess urinary symptoms, such as incomplete emptying, frequency, urgency, and weak stream. Each question has six possible answers, ranging from 0 to 5 points, with higher numbers indicating more severe symptoms.
Change in Male Sexual Health Questionnaire Short-Form (MSHQ-EjD-SF) | Baseline, 6 weeks, 15 weeks
  The Male Sexual Health Questionnaire Short-Form (MSHQ-EjD-SF) is a 4 item questionnaire to assess the degree of ejaculatory dysfunction in men. The domains include three ejaculatory function items and one ejaculation bother item.
Change in Quality of Life Scale | Baseline, 6 weeks, 15 weeks
  The Quality of Life Scale is a 16-item instrument that measures six domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, recreation, and independence on a scale of 1 to 7 where a low value indicates "terrible" and a high value indicates "delighted". Higher overall scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R Humphreys, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials